CLINICAL TRIAL: NCT06497335
Title: Accuracy of Non Invasive Hemoglobin Measure by SpHb Device in Post Operative Anemia Diagnosis: a Validation Study in Gynecological Surgery Department of Angers 's University Hospital
Brief Title: Accuracy of Non Invasive Hemoglobin Measure by SpHb Device in Post Operative Anemia Diagnosis
Acronym: SpHb_gyneco
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 24_0206
Record Dates: First submitted 2024-06-18; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Anemia
Keywords: post operative screening; anemia; iron deficiency; diagnosis
MeSH Terms: conditions — Anemia; Iron Deficiencies; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: non invasive hemoglobin measure — non invasive hemoglobin measure

SUMMARY:
Non invasive Hemoglobin monitoring by SpHb device had been developed to assess Hemoglobin level during hemorrhagic surgery. It's accuracy to detect post operative anemia on a single post operative measure has been recently demonstrated on a cohort of post operative orthopedic patient and it's routine use has been generalized to other surgical department. This study aims to valid these finding on a cohort of post operative patients from gynaecological department.

ELIGIBILITY:
Inclusion Criteria:

* being hospitalized for gynecological procedure: hysterectomy or cancer related annexectomy
* > 18 years

Exclusion Criteria:

* non french speaker
* being under a legal individual protection measure
* not being able to consent
* being opposed to data collection

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: population of gynecological surgical department
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
accuracy between SpHb measure and Hemoglobin level on the post operative blood sample | at 2 and 8 months after establishment of PBM protocol
  level of immediate post operative SpHb measure compared to blood hemoglobin measure, ROC curve

SECONDARY OUTCOMES:
Spearman correlation coefficient | at 2 and 8 months after establishment of PBM protocol
  correlation between Laboratory Hb and SpHb measure
Kappa coefficient | at 2 and 8 months after establishment of PBM protocol
  correlation between SpHb measure and correct classification of patients anemia vs no anemia
Intra class correlation coefficient | at 2 and 8 months after establishment of PBM protocol
  correlation between Laboratory measurement and SpHb measurement
Subgroup analysis of ROC curve (classes of age 18-30; 30-40; 40-50; >50) | at 2 and 8 months after establishment of PBM protocol
  comparison of ROC curve areas in subgroups
impact of body temperature on accuracy of SpHb | at 2 and 8 months after establishment of PBM protocol
  comparison of ROC curve areas in subgroups of temperature (classes of temperature : <35; 35-36; >36)
impact of perfusion index on accuracy of SpHb | at 2 and 8 months after establishment of PBM protocol
  comparison of ROC curve areas in subgroups of perfusion index (good or low perfusion index)
impact of leght between SpHb measurement and laboratory Hb measurement on accuracy | at 2 and 8 months after establishment of PBM protocol
  comparison of ROC curve areas in subgroups of lenght in days between SpHb measurement and Laboratory Hb measurement

CONTACTS AND LOCATIONS:
Overall Officials: Sigismond Lasocki, Principal Investigator — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: No